CLINICAL TRIAL: NCT03199274
Title: Ultrasound Microbubble Destruction and Perfusion Quantification for Improving Radioembolization Therapy of Hepatocellular Carcinoma
Brief Title: Perflutren Protein-Type A Microspheres and Contrast-Enhanced Ultrasound in Improving Response to Radioembolization Therapy in Patients With Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, john eisenbrey, Associate Professor of Radiology, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17F.222; 5R01CA238241 (NIH); JT 10205 (Other: JeffTrial Number)
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — FS 069

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (perflutren protein-type A microspheres, CEUS) (Experimental): Patients receive perflutren protein-type A microspheres IV over 10 minutes and undergo CEUS over 60 minutes at 1-6 hours and at approximately 7 and 14 days after yttrium Y-90 radioembolization.
  Interventions: Procedure: Yttrium-90 Microsphere Radioembolization; Drug: Perflutren Protein-Type A Microspheres; Procedure: Dynamic Contrast-Enhanced Ultrasound Imaging
- Group II (standard of care) (Active Comparator): Patients undergo standard of care yttrium Y-90 radioembolization.
  Interventions: Procedure: Yttrium-90 Microsphere Radioembolization

INTERVENTIONS:
Procedure: Yttrium-90 Microsphere Radioembolization — Undergo standard of care Y-90 radioembolization
  Other Names: Yttrium Y 90 Microsphere Therapy; Yttrium-90 Radioembolization
Drug: Perflutren Protein-Type A Microspheres — Given IV.
  Other Names: Optison
  Arms: Group I (perflutren protein-type A microspheres, CEUS)
Procedure: Dynamic Contrast-Enhanced Ultrasound Imaging — Undergo CEUS
  Arms: Group I (perflutren protein-type A microspheres, CEUS)

SUMMARY:
This phase II trial studies how well perflutren protein-type A microspheres and contrast-enhanced ultrasound work in improving response to radioembolization therapy in patients with liver cancer. Ultrasound contrast agents, such as perflutren protein-type A microspheres, use gas microbubbles to improve image quality. Using contrast-enhanced ultrasound imaging will "pop" these microbubbles and cause tumors to become more sensitive to radiation therapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Characterize the ability of localized ultrasound contrast agent destruction to improve hepatocellular carcinoma (HCC) response to yttrium Y-90 (Y90) radioembolization.

SECONDARY OBJECTIVE:

I. Determine if contrast-enhanced ultrasound estimated tumor perfusion can reliably predict HCC response to radioembolization 1-14 days post treatment.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive perflutren protein-type A microspheres intravenously (IV) over 10 minutes and undergo contrast-enhanced ultrasound (CEUS) over 60 minutes at 1-6 hours and at approximately 7 and 14 days after yttrium Y-90 radioembolization.

GROUP II: Patients undergo standard of care yttrium Y-90 radioembolization.

After completion of study treatment, patients are followed up at 1 month and at 3-4 months.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for sub-lobar radioembolization therapy of a previously untreated HCC mass < 6 cm visible on grayscale ultrasound
* Be medically stable
* If a female of child-bearing age, have a negative pregnancy test prior to each ultrasound exam
* Have signed informed consent to participate in the study

Exclusion Criteria:

* Females who are pregnant or nursing
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable; for example:

  * Patients on life support or in a critical care unit
  * Patients with unstable occlusive disease (e.g., crescendo angina)
  * Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia
  * Patients with uncontrolled congestive heart failure (New York heart Association [NYHA] class IV)
* Patients with recent cerebral hemorrhage
* Patients with known sensitivities to albumin, blood, or blood products
* Patients with known hypersensitivity to perflutren
* Patients with known cardiac shunts
* Patients with known congenital heart defects
* Patients with severe emphysema, pulmonary vasculitis, or a history of pulmonary embolism
* Patients with respiratory distress syndrome
* Patients with a history of bleeding disorders
* Patients with bilirubin levels > 2 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Eisenbrey, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Wessner CE, Forsberg F, Lyshchik A, O'Kane P, Bradigan K, Liu JB, Delaney LJ, Anton K, Topper SR, Civan J, Maley W, Keith SW, Shaw CM, Eisenbrey JR. Microbubble-based Radiosensitization of Hepatocellular Carcinoma: Evaluation of Safety and Efficacy in a Phase II Randomized Trial. Radiology. 2025 Sep;316(3):e250083. doi: 10.1148/radiol.250083. PMID 41025990
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (Perflutren Protein-type A Microspheres, CEUS) | Group II (Standard of Care)
Started | 52 | 52
Completed | 48 | 50
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Deemed screen fail because he had no arteries to access during flow study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Perflutren Protein-type A Microspheres, CEUS) | Group II (Standard of Care) | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 36 | 38 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 8 | 28
  Male | 32 | 44 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 50 | 50 | 100
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 37 | 38 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response to Yttrium Y-90 Radioembolization
Description: Measured using the modified Response Evaluation Criteria in Solid Tumors. Will be tested with a non-parametric Mann- Whitney U-test of the difference in response distributions between control (radioembolization alone) and experimental group (ultrasound-triggered microbubble destruction [UTMD] + radioembolization). The outcome variable in this analysis, the modified Response Evaluation Criteria in Solid Tumors (mRECIST) score, is treated as an ordinal variable in this analysis. Tumor response assessed using modified Response Evaluation Criteria in Solid Tumors (mRECIST). The mRECIST scale includes four ordered categories:
  * Complete Response (best outcome)
  * Partial Response
  * Stable Disease
  * Progressive Disease (worst outcome)
Time Frame: Up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Perflutren Protein-type A Microspheres, CEUS) | Group II (Standard of Care)
Number analyzed (Participants) | 48 | 50
Participants
  Stable Disease | 2 | 17
  Partial Response | 17 | 17
  Complete Response | 25 | 13
  Progressive Disease | 4 | 3

2. Primary Outcome: Tumor Perfusion Measured by Contrast-enhanced Ultrasound Between Ultrasound-triggered Microbubble Destruction Pulses
Description: Perfusion will be characterized in terms of contrast replenishment time intensity curves fit with a 2-parameter exponential recovery curve. The relationship between the normalized perfusion values from this image processing and the patients' subsequent mRECIST scores in the UTMD + radioembolization group will be evaluated with Spearman's rank order correlation. Tumor perfusion measured as fractional vascularity (%) using contrast-enhanced ultrasound (CEUS). Values range from 0% (no perfusion) to 100% (maximal perfusion).
Time Frame: Up to 14 days
Population: Contrast-enhanced ultrasound (study intervention) is only collected from patients in Arm 1.
Measure: Mean (Standard Deviation); unit: percentage of tumor vascularity
Groups:
- Group II (Standard of Care): Patients undergo standard of care yttrium Y-90 radioembolization. Yttrium-90 Microsphere Radioembolization: Undergo standard of care Y-90 radioembolization
Arm/Group | Group I (Perflutren Protein-type A Microspheres, CEUS) | Group II (Standard of Care)
Number analyzed (Participants) | 48 | 0
percentage of tumor vascularity
  Viable Tumors | 62 (28) |
  Non-Viable Tumors | 38 (24) |

ADVERSE EVENTS:
Time Frame: From enrollment through 3-4 months post-treatment
Description: Adverse events were assessed through participant reports, systematic review of medical records, and clinical monitoring at 1 month and 3-4 month follow up visits
Arm/Group | Group I (Perflutren Protein-type A Microspheres, CEUS) | Group II (Standard of Care)
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 4/52 | 2/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (Perflutren Protein-type A Microspheres, CEUS) (N=52) | Group II (Standard of Care) (N=52)
Fever (General disorders) | 4 | 0
Hives/rash (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Possible Seizure (Nervous system disorders) | 0 | 1
Dyspnea (General disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Shoulder Pain (General disorders) | 1 | 0
Shortness of Breath (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT03199274/Prot_SAP_000.pdf